CLINICAL TRIAL: NCT02866344
Title: Prospective Randomized Comparison of Resection and Microwave Ablation for Resectable Colorectal Cancer Liver Metastases
Brief Title: Resection Versus Microwave Ablation for Resectable Colorectal Cancer Liver Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00083181; 06-16-02A (Other: Atrium)
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Hepatic Neoplasms
Keywords: Microwave ablation; Ablation techniques; Operative surgical procedures; Hepatic resection; Surgery; Outcomes assessment
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Liver Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave ablation (Experimental): Patients will be given general anesthesia. A laparoscopic trocar and additional ports will be placed under direct visualization and pneumoperitoneum will be established. Once the operating surgeon determines that the lesions as evaluated on intraoperative ultrasound remain amenable to MWA, ablations will be performed with a 2.45-gigahertz (GHz) generator with a 1.8-mm-diameter transcutaneous antenna (Acculis pMTA Accu2i; AngioDynamics Inc., Denmead, Hampshire, UK). Additional ablations will be performed sequentially. Laparoscopic core needle biopsy of lesions will be performed and submitted for permanent pathologic sectioning per current treatment standards. At the conclusion of the ablation, a collapsed titanium clip will be inserted into the microwave antenna tract as a radiographic fiducial marker. Hemostasis of the ablation track will be ensured using a combination of microwave energy, monopolar electrocautery, and/or topical hemostatics.
  Interventions: Procedure: Microwave ablation
- Hepatic resection (Active Comparator): General anesthesia will be induced. A laparoscopic trocar and additional ports will be placed under direct visualization and pneumoperitoneum will be established. The liver will be evaluated with intraoperative ultrasound (BK Medical A/S, Herlev, Denmark). Laparoscopic core needle biopsy of lesions will be performed. Partial hepatectomy may be carried out with parenchymal precoagulation with radiofrequency electrosurgical devices such as the LigaSure™ (Covidien, Medtronic; Minneapolis, MN), Harmonic® (Ethicon Endosurgery; Cincinnati, OH), or saline-coupled radiofrequency ablation device (Aquamantys™; Covidien/Medtronic; Minneapolis, MN); hepatic parenchymal transection can be performed as above or with the use of stapling devices to ligate and divide parenchyma. Hepatic vascular inflow occlusion will be performed at the surgeon's discretion. A topical hemostatic may be used along the transected hepatic parenchyma. Resected specimens will be preserved in formalin for pathology.
  Interventions: Procedure: Hepatic resection

INTERVENTIONS:
Procedure: Microwave ablation — Laparoscopic or robot-assisted laparoscopic microwave ablation of cancerous lesions with a 2.45-GHz microwave generator and a 1.8-mm-diameter transcutaneous antenna.
  Arms: Microwave ablation
Procedure: Hepatic resection — Laparoscopic or robot-assisted laparoscopic surgical resection of cancerous lesions.
  Other Names: Surgery
  Arms: Hepatic resection

SUMMARY:
This single-center, prospective, randomized clinical trial is designed to compare the clinical characteristics and outcomes of hepatic resection and microwave ablation (MWA) to determine the optimal operative intervention for the local treatment of resectable colorectal cancer liver metastases. The primary aim of this study is to test the following hypothesis: 2-year local disease control is equivalent between patients receiving the experimental therapy (MWA) and patients receiving the standard therapy (hepatic resection) as treatment for colorectal cancer liver metastases determined to be resectable by radiographic imaging. Secondarily, the investigators expect that 2-year intrahepatic (regional) and metastatic disease recurrence rates are equivalent between the two treatment arms in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the colon or rectum (diagnosed at the time of colon or rectal resection or on endoscopic biopsy) with liver metastases (by liver biopsy or by history of biopsy-proven colon/rectal cancer with characteristic imaging findings):
* Imaging showing typical features of colorectal cancer liver metastasis;
* Cytologic/histologic diagnosis of colorectal cancer or colorectal cancer liver metastasis.
* No more than 3 hepatic metastatic lesions noted on preoperative imaging
* No lesion greater than 5 cm in maximal dimension
* Adequate clinical condition to undergo laparoscopic or robot-assisted laparoscopic liver resection or microwave ablation as treatment for colorectal cancer liver metastases
* Willing and able to give informed consent

Exclusion Criteria:

* Radiologic (computed tomography or magnetic resonance imaging) evidence of invasion into major portal/hepatic venous branches and no extrahepatic metastases
* Evidence of recurrent disease adjacent to a previous ablation or resection site
* Severe renal dysfunction (creatinine clearance of <40 mL/min)
* Pregnant or nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Local disease control at the site of intervention | 2 years
  Local disease control is measured from time of randomization and is defined as the absence of local recurrence of metastatic adenocarcinoma of the colon or rectum as determined by diagnostic imaging.

SECONDARY OUTCOMES:
Overall survival | 1, 2, 3, 5 years
Intrahepatic disease-free survival | 1, 2, 3, 5 years
Postoperative morbidity | 1 month and 3 months
Postoperative mortality | 1 month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dionisios Vrochides, MD PhD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided